CLINICAL TRIAL: NCT03096587
Title: Effect Of Using XP Endo Finisher Versus Ultrasonic Activated Irrigation On Post-operative Pain In Single Visit Endodontic Treatment of Teeth With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: Effect Of XP Endo Finisher Versus Ultrasonic Activated Irrigation On Post-operative Pain In Endodontic Treatment of Symptomatic Irreversible Pulpitis
Acronym: RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nouran Ahmed Hany Asal, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBC-CU-2017-03-19
Record Dates: First submitted 2017-03-25; First posted 2017-03-30 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: XP Endo Finisher; ultrasonic activated irrigation; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Masking Description: The patient will be blinded and will not know the group he is in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- XP Endo Finisher file (Experimental): XP Endo Finisher file is used to activate irrigation as a final step in irrigation protocol
  Interventions: Device: XP Endo Finisher
- ultrasonic activated irrigation (Active Comparator): ultrasonic activated irrigation as a final step in irrigation protocol
  Interventions: Device: ultrasonic activated irrigation

INTERVENTIONS:
Device: XP Endo Finisher — a flexible single use NiTi file with small diameter and no taper, changes from straight M-phase to A-phase in body temperature
  Arms: XP Endo Finisher file
Device: ultrasonic activated irrigation — by Satelec,Acteon, France
  Other Names: Irrisafe
  Arms: ultrasonic activated irrigation

SUMMARY:
Recruited patients with symptomatic irreversible pulpitis are assigned to interventional (XP Endo Finisher file) and control group(ultrasonic activated irrigation) to undergo single visit endodontic treatment and record postoperative pain afterwards.

DETAILED DESCRIPTION:
The investigator will recruit patients from the clinic of endodontics in faculty of oral and dental medicine, Cairo university.

The patients who are found eligible to the criteria, will be randomly assigned to either the control group (ultrasonic activated irrigation )or to the intervention group( XP Endo-Finisher file). Endodontic treatment will be done in single visit.

After the visit, patients will be asked to record post operative pain by NRS (Numerical Rate Scale)in a given sheet.

ELIGIBILITY:
Inclusion Criteria:

1. Medically- free of any systemic disease
2. Male or female
3. Patients with age range 25-45
4. Symptomatic irreversible pulpitis in single rooted single canal teeth without apical periodontitis.
5. Teeth with mature root
6. Restorable teeth
7. Teeth without calcified root canals
8. Teeth without root caries
9. Teeth without internal or external root resorption
10. Teeth with no sign of crack formation
11. Teeth without anatomic abnormalities

Exclusion Criteria:

1. Pregnant females.
2. If analgesics have been administrated during the past two weeks preoperatively.
3. Patients having bruxism or clenching.
4. Multi rooted or multi canaled teeth.
5. Patients with swelling or acute peri-apical abscess.
6. Previously endodontically treated teeth
7. periodontally affected teeth .

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-04-15 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
post-operative pain | up to 1 week after the visit
  measured by NRS (Numerical rate scale)

SECONDARY OUTCOMES:
Number of taken analgesic tablets | within a week after the visit
  counted by the patient and recorded in a given chart

CONTACTS AND LOCATIONS:
Overall Officials: Nouran A Hany, BDS, Principal Investigator — Department of endodontics -Faculty of Oral and Dental Medicine-Cairo university; Shaimaa I Gawdat, PHD, Study Director — Department of endodontics -Faculty of Oral and Dental Medicine-Cairo university; Hebatallah M El-Far, Professor, Study Chair — Department of endodontics -Faculty of Oral and Dental Medicine-Cairo university
Locations (1):
- Faculty of Oral and dental medicine, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Alves FR, Andrade-Junior CV, Marceliano-Alves MF, Perez AR, Rocas IN, Versiani MA, Sousa-Neto MD, Provenzano JC, Siqueira JF Jr. Adjunctive Steps for Disinfection of the Mandibular Molar Root Canal System: A Correlative Bacteriologic, Micro-Computed Tomography, and Cryopulverization Approach. J Endod. 2016 Nov;42(11):1667-1672. doi: 10.1016/j.joen.2016.08.003. Epub 2016 Sep 15. PMID 27641947
- [Result] Middha M, Sangwan P, Tewari S, Duhan J. Effect of continuous ultrasonic irrigation on postoperative pain in mandibular molars with nonvital pulps: a randomized clinical trial. Int Endod J. 2017 Jun;50(6):522-530. doi: 10.1111/iej.12666. Epub 2016 Jun 28. PMID 27248848
- [Result] Sadaf D, Ahmad MZ. Factors associated with postoperative pain in endodontic therapy. Int J Biomed Sci. 2014 Dec;10(4):243-7. PMID 25598754